CLINICAL TRIAL: NCT06510725
Title: Effect of Multitarget Transcranial Direct Current Stimulation (tDCS) in Patients With Neuropathic Pain
Brief Title: Effect of Multitarget tDCS for Neuropathic Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Beijing Tiantan Hospital (Other); Second Affiliated Hospital of Tsinghua University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: zhuhongwei
Record Dates: First submitted 2024-07-09; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mutitarget tDCS (Experimental): Subjects will receive 20 minutes of active transcranial direct current stimulation at 2mA applied to DLPFC and M1 alternately for ten consecutive weekdays, with each target stimulated for 5 sessions.
  Interventions: Device: Mutitarget tDCS
- Single-target tDCS (Experimental): Subjects will receive 20 minutes of active transcranial direct current stimulation at 2mA applied to M1 for ten consecutive weekdays.
  Interventions: Device: Single-target tDCS
- Sham tDCS (Sham Comparator): Subjects will receive 20 minutes of sham transcranial direct current stimulation. Ramps up and down will be applied for 15 seconds each at the beginning and end of the session. The current will be 0 mA during the interval between the initial and final ramps. Subjects will undergo stimulation once a day for ten consecutive weekdays.
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Mutitarget tDCS — Subjects will receive 20 minutes of active transcranial direct current stimulation at 2mA applied to DLPFC and M1 alternately for ten consecutive weekdays, with each target stimulated for 5 sessions.
  Arms: Mutitarget tDCS
Device: Single-target tDCS — Subjects will receive 20 minutes of active transcranial direct current stimulation at 2mA applied to M1 for ten consecutive weekdays.
  Arms: Single-target tDCS
Device: Sham tDCS — Subjects will receive 20 minutes of sham transcranial direct current stimulation. Ramps up and down will be applied for 15 seconds each at the beginning and end of the session. The current will be 0 mA during the interval between the initial and final ramps. Subjects will undergo stimulation once a day for ten consecutive weekdays.
  Arms: Sham tDCS

SUMMARY:
This study aims to conduct a randomized controlled trial to evaluate the effect of multitarget transcranial direct current stimulation (tDCS) on pain, depression, anxiety, quality of life and sleep, in patients with neuropathic pain.

DETAILED DESCRIPTION:
The present multicenter, randomized, double-blind, sham-controlled, parallel-group trial aims to evaluate the effect of multitarget transcranial direct current stimulation (tDCS) in patients with neuropathic pain.

The patients will be randomized to receive one of 3 treatment arms: multitarget stimulation, single-target stimulation and sham stimulation. All patients received 20 minutes of active or sham tDCS once a day for 10 consecutive weekdays. In multitarget group, subjects will receive 2mA tDCS applied to M1 and DLPFC alternately, with each target stimulated for 5 sessions. In single-target group, 2mA tDCS will target M1 only. In sham group, subjects will receive sham tDCS. Ramps up and down will be applied for 15 seconds each at the beginning and end of the session. The current will be 0 mA during the interval between the initial and final ramps.

ELIGIBILITY:
Inclusion Criteria:

1. Female or males aged between 18 and 75 years.
2. Pain fulfilling the criteria for probable or definite neuropathic pain and scoring ≥4/10 at Douleur Neuropathique 4 Questions.
3. Pain duration of at least 3 months and average pain intensity scoring ≥4/10 at Numeric Rating Scale.
4. Stable pharmacological treatment for at least 4 weeks prior to the study and throughout the trial.
5. Informed consent obtained.

Exclusion Criteria:

1. Pregnancy or lactation.
2. Active central nervous system diseases including but not limited to brain tumour, intracranial hypertension, past or current epilepsy.
3. Unable to complete the questionnaire due to language abilities or reduced cognitive functioning.
4. Alcohol or substance abuse.
5. Common contraindications for transcranial direct current stimulation including but not limited to skull defect, implanted device or metal in the brain, severe cardiopulmonary, renal or hepatic diseases.
6. Unwilling to comply with the treatment or follow-up assessments.
7. Participating in another clinical trial within 3 months prior to enrollment of this clinical trial.
8. Any patient deemed unsuitable for enrollment by the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in average pain intensity | from baseline to week 2
  Change in average pain intensity from baseline to week 2, average pain intensity corresponds to average pain over the last 24 hours on the Brief Pain Inventory

SECONDARY OUTCOMES:
Change in Brief Pain Inventory (BPI): Average pain over the last 24 hours | from baseline to week 6 and week 10
Change in BPI: Maximal pain over the last 24 hours | from baseline to week 2, week 6 and week 10
Change in BPI: Minimal pain over the last 24 hours | from baseline to week 2, week 6 and week 10
Change in Neuropathic Pain Symptoms Inventory (NPSI): Burning pain | from baseline to week 2, week 6 and week 10
Change in NPSI: Deep pain | from baseline to week 2, week 6 and week 10
Change in NPSI: Paroxysmal pain | from baseline to week 2, week 6 and week 10
Change in NPSI: Evoked pain | from baseline to week 2, week 6 and week 10
Change in NPSI: Paraesthesia | from baseline to week 2, week 6 and week 10
Change in Hamilton Depression Scale (HAMD) | from baseline to week 2, week 6 and week 10
Change in Hamilton Anxiety Scale (HAMA) | from baseline to week 2, week 6 and week 10
Change in Pittsburgh sleep quality index (PSQI) | from baseline to week 6 and week 10
Change in five-level EuroQol five-dimensional questionnaire (EQ-5D-5L): EQ-VAS | from baseline to week 2, week 6 and week 10
Change in EQ-5D-5L: Utility score | from baseline to week 2, week 6 and week 10
Proportion of participants with meaningful improvement compared with baseline (score as 1 or 2) in Patient Global Impression of Change (PGIC) | Week 2, Week 6, Week 10
  PGIC includes 7 ranks ranging from 1 to7 (1= very much improved; 2= moderately improved; 3=slightly improved; 4= no change; 5= slightly worsened; 6= moderately worsened; 7= very much worsened)

IPD SHARING:
Plan to Share IPD: No